CLINICAL TRIAL: NCT03992469
Title: Study to Evaluate Safety, Tolerability, and Early Efficacy of Oral E-B-FAHF-2 in Subjects With Mild-To-Moderate Crohn's Disease
Brief Title: Study to Evaluate Safety, Tolerability and Efficacy of Oral E-B-FAHF-2 in Mild-to-Moderate Crohn's Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Dunkin, Assistant Professor, Pediatrics, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 19-0125; 0266-3308 (Other Grant/Funding Number: The Helmsley Charitable Trust)
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Crohn's Disease
Keywords: Entocort EC induction; double blind, controlled safety/tolerability trial; open label exploratory efficacy trial; mild-to-moderate crohn's disease; Chinese Herbal Therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Safety and Tolerability phase is a double blind randomized controlled trial to evaluate safety and tolerability over 8 weeks. This is followed by an open-labeled exploratory efficacy extension phase for 6 months.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind placebo controlled safety trial with random assignment to groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-B-FAHF-2 (Experimental): Low dose EBFAHF-2 (29 mg/kg/d divided two times a day) for 2 weeks followed by a full dose (71mg/kg/d divided two times a day) for 6 weeks
  Interventions: Drug: EBFAHF-2
- Placebo (Placebo Comparator): capsules are identical in appearance to EBFAHF-2 capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EBFAHF-2 — EBFAHF-2 is a 0.55g capsule that is easy to swallow. The quality, safety and consistency of EBFAHF-2 are established per FDA guidance under a botanical drug title. Low dose (maximum of 2 capsules bid) and full dose (maximum of 5 capsules bid). Weight based dosing will ensure an equivalent amount is given to each individual.
  Arms: E-B-FAHF-2
Drug: Placebo — Placebo capsules made of cornstarch
  Arms: Placebo

SUMMARY:
Crohn's disease (CD) is the major form of inflammatory bowel disease (IBD) affecting adults. It is a life-long disease characterized by chronic and relapsing inflammation of the gastrointestinal tract. CD has multiple clinical phenotypes and disease severities that determine which therapy the study team utilizes. Currently, there are numerous treatment options for subjects with moderate-severe CD, but few that are approved to treat and maintain remission for the one-third of patients who present with mild-to-moderate disease. The study team hypothesizes that Butanol Purified Food Allergy Herbal Formula-2 (B-FAHF-2) will be safe and effective for maintaining remission of mild-to-moderate CD and can fill this therapeutic void. CD affects 241 per 100,000 adults in the United States and the incidence in both adults and children has increased in the past 60 years. One such potential therapy is Food Allergy Herbal Formula-2 (FAHF-2) which was originally developed to treat food allergy and has received FDA investigational new drug approval under the botanical drug title for treating patients with multiple food allergies. A completed phase I study showed that FAHF-2 is safe and well tolerated. A Phase II trial revealed that a high pill burden with FAHF-2 caused poor compliance. A butanol purified form of FAHF-2 (B-FAHF-2) is a more concentrated form of FAHF-2 which has also received an IND (FDA IND#77,468) and reduces the pill burden and improves compliance. Interestingly, the herbal components in B-FAHF-2 have long been used in Traditional Chinese Medicine (TCM) to treat gastrointestinal disorders including colitis. The study team has shown that B-FAHF-2 non-toxically inhibits TNF-#, a major inflammatory cytokine involved in CD, as well as multiple other pro-inflammatory cytokines produced by human peripheral blood mononuclear cells (PBMCs) and intestinal mucosa from subjects with CD. In addition, the study team has shown that FAHF-2 prevents disease progression in a murine model of colitis. The study team hypothesizes that E-B-FAHF-2 will be safe and effective for treating mild-to-moderate CD and can fill this therapeutic void. The study team proposes to investigate the safety and tolerability of B-FAHF-2 in subjects with mild-to-moderate CD. The goal is to establish safety and tolerability and explore efficacy at maintaining remission in this select patient population. Importantly, the study team will also determine the immunotherapeutic effects of E-B-FAHF-2 on PBMCs and intestinal mucosa to determine if there are immunologic alterations that would indicate that controlled efficacy evaluations of E-B-FAHF-2 are warranted. The new IND number is 143453. The FDA has completed their safety review of this protocol and has concluded that the study team's clinical trial may proceed with the proposed clinical investigation for Crohn's disease.

DETAILED DESCRIPTION:
The study team's current proposed study uses the same investigational agent, E-B-FAHF-2, being studied for food allergy under an active IND, and seeks to determine if this formula is safe for the treatment of mild-to-moderate CD. The study team's major goal focuses on safety, tolerability, beneficial immunomodulatory effect, and preliminary clinical efficacy of B-FAHF-2 to maintain remission in subjects with mild-to-moderate CD. B-FAHF-2 is currently undergoing a phase II clinical trial for treatment of food allergy, thus increasing the ease of obtaining an FDA IND for B-FAHF-2 use in CD. Preliminary data were generated in the study team's ongoing FAHF-2 and B-FAHF-2 studies on food allergy and IBD. In developing a botanical drug from a traditional Chinese medicine (TCM) formula, standardization of product is key to ensure safety, consistency, and potency. An IND for B-FAHF-2 has been accepted by the FDA, and is documented that the product's quality, safety and standardized methodology have been demonstrated. To date, the study team has demonstrated the safety of B-FAHF-2 in animal models and the safety and tolerability of B-FAHF-2 in patients, including adults and children with food allergy. The most specific data relevant to this proposal are the suppression by FAHF-2/B-FAHF-2 of TNF-alpha production by PBMC's and intestinal specimens from children with CD and the abrogation of colitis in a murine model.

CD is a life-long chronic, relapsing, immune mediated inflammatory disease characterized by inflammation in the gastrointestinal tract. Treatment is aimed at controlling mucosal inflammation, and thus symptoms of the disease, by inducing and then maintaining remission. Since CD causes abdominal pain, decreased appetite, malabsorption and diarrhea, children are particularly vulnerable because inadequate nutrition can lead to potentially irreversible growth stunting and delayed maturity. There is a lack of maintenance therapies for children and adults with mild-to-moderate disease since many of the medications used to treat CD. including steroids, immunomodulators and biological therapies are geared towards treating moderate-to-severe disease. The most commonly used medications for treatment and maintenance of remission in mild-to-moderate CD are 5-ASA compounds and antibiotics but they are not FDA approved and the literature does not support their utility in CD. Based on the inhibition of TNF-alpha by B-FAHF-2 and FAHF-2 in vitro, the study team hypothesizes that E-B-FAHF-2 will be safe and effective therapy that will fill this therapeutic void. The study team proposes to test the safety and tolerability of E-B-FAHF-2 in subjects with recently diagnosed mild-to-moderate CD that responds to induction with Entocort EC. To minimize any potential risk by exposing a large number of subjects to treatment: the study team will conduct the study in subjects 18-30 years old to assess for safety, tolerability and determine immunological and/or efficacy signals (subjective and objective measures). Since E-B-FAHF-2 is likely to be slow to work, subjects will be induced with Entocort EC for 8 weeks. Responders will then be enrolled in the trial. The safety and tolerability trial is eight weeks long, double blind, placebo controlled dose escalation trial of E-B-FAHF-2 in subjects who responded to induction therapy with Entocort EC. This portion of the study will serve to ensure safety and tolerability of E-B-FAHF-2. Subjects will be seen every 2 weeks and contacted by phone in between study visits to assess for any adverse events (AEs). This will be followed by a 6 month long, open-label exploratory extension trial of E-B-FAHF-2 monotherapy to ensure the sub-chronic safety as well as determine of there is any efficacy or immunologic alteration to pursue in randomized efficacy trials. During this phase, subjects will have follow-up visits every 4 weeks to assess for AEs and efficacy outcomes. In addition, a subset of 4 subjects will participate in PK studies for one of the visits during this phase. The exploratory efficacy phase of the study will be conducted in a population of subjects naive to immunomodulators, systemic steroids and biologics. This study population will provide us with an opportunity to determine the safety and immunologic effects of E-B-FAHF-2 in CD without the interference of systemic immunomodulating medications.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfill all of the following criteria to be eligible for inclusion in the study:

* Male and female subjects with Crohn's disease (CD), 18-60 years of age and otherwise in good health as determined by medical history and physical examination
* Subjects weighing 25kg or more
* History of ileal or ileal-colonic CD that is mild-to-moderate in severity as determined by standard history, physical, endoscopy scoring results, CD Activity Index (CDAI); patients with severe disease, which can be rapidly progressive and result in gastrointestinal hemorrhage, intestinal fistulas, abscesses and other complications, will be excluded because their risk of requiring rescue medications including steroids and biologicals as well as hospitalization or surgery are high.
* The subject is able to swallow the required capsules and tablets.
* The subject has been immunized according to the guidelines set forth by the CDC.
* The subject agrees to participate in the study.
* Females of childbearing potential must be sexually inactive or take effective birth control measures, as deemed appropriate by the investigator, for the duration of the study.
* Evidence of inflammation on colonoscopy with an SES-CD >3.
* Either an elevated fecal calprotectin or an elevated CRP.
* Willing and able to undergo upper endoscopy and colonoscopy with disease flares and after 6 months of treatment for the assessment of disease as per the standard of care for CD.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Subjects will be excluded from the study if any of the following apply:

* Patients with severe disease as determined by CDAI, or SES-CD scores at initial endoscopy of greater than 16, or strictures or large ulcerations on endoscopy that exemplify severe disease.
* Acute febrile illness within 1 week before administration of study therapeutic formula.
* Any history of other systemic diseases that, in the investigator's opinion, would preclude the subject from participating in this study, e.g. other autoimmune disease, neoplasm, HIV or hepatitis infection.
* Abnormal hepatic function (ALT, AST or bilirubin >2 x upper limit of normal).
* Abnormal bone marrow function (WBC <4 x 103/mm3; platelets <100 x 103/mm3).
* Abnormal renal function (BUN and creatinine >1.5 x upper limit of normal for age or abnormal eGFR for age and race).
* Clinically significant abnormal electrocardiogram.
* Participation in another experimental therapy study within 30 days of this study.
* History of alcohol or drug abuse.
* Pregnant or lactating female subjects: females of childbearing potential will need a negative pregnancy test at screening and at each visit to be considered and continued in this study. Lactating females will be excluded from the study.
* Active perirectal disease including fistuli or abcesses.
* Use of any other CAM products.
* Known allergy to FAHF-2/B-FAHF-2 or any of its components.
* Concurrent use of any medications known to alter CYP3A function.
* Any other medical concerns not listed above that in the invistigator's opinion may pose additional risks, interfere with adherence, or impact the quality or interpretation of the data.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Number of grades of adverse events | 8 months
  Safety and tolerance will be assessed by number of adverse events using a previously established grading system by the study team.

SECONDARY OUTCOMES:
Number of participants requiring an escalation in therapy. | 6 months
  Before enrollment and at each visit a CDAI will be assessed. The CDAI is a clinical score for adults that includes history items, physical examination items, and laboratory tests and is based on the past 7 days. A score of <150 is defined as remission, 151-219 as mild activity, 220-450 as moderate activity and >450 as severe activity. Clinical response is defined as a decrease in score of at least 70 points or >25% in subjects with baseline CDAI >220.
  Any escalations in therapy will be recorded and assessed as described above.
Fecal Calprotectin | 6 months
  The level of calprotectin in stool as a way to detect inflammation in the intestines.
PROMIS Profile 29 | 6 months
  PROMIS Profile-29 is a validated, self-report collection of 4-item short forms that uses a 5-point Likert scale to assess anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities. PROMIS measures are scored on the T-score metric. High scores mean more of the concept being measured. Norm-based scores have been calculated for each domain on the PROMIS measures, so that a score of 50 represents the mean or average of the reference population. A score of 60 means that the person is one standard deviation above the reference population(standard deviation=10).
Self Efficacy Scale: IBDSES | 6 months
  This self-administered efficacy scale includes 13 items that assess how patients with IBD manage items related to their disease and everyday life. The validated scale uses 5-point Likert scales for each item. the total score ranges from 13 to 65 with a lower score indicating lower self-efficacy.
Immunologic Changes in PBMC cytokine levels | 6 months
  PBMCs will be obtained along with routine labs at the start of the safety trial and after starting (week 8), during (week 12 and 20) and completing the exploratory extension trial (week 32).

CONTACTS AND LOCATIONS:
Overall Officials: David Dunkin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.Any purpose.Data are available indefinitely at (Link to be included).
URL: https://vivli.org/

REFERENCES:
- Available data/document: Individual Participant Data Set — https://vivli.org/